CLINICAL TRIAL: NCT03939286
Title: Multimodal Imaging Study on Physical Activity in Patients With Alzheimer's Disease
Acronym: DEMENTIA-MOVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19-064
Record Dates: First submitted 2019-04-05; First posted 2019-05-06 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Neuropsychological Tests; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: In total, about 50 study participants will be examined in a prodromal or symptomatic early stage of Alzheimer's disease. These should be distributed equally randomized into two groups: a movement group (n = 25) with intensified training (equipment, coordination, balance) and a control group with continuation of physical activity as usual and participation in a psychoeducational program (n = 25).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- movement group (Other): intensified training (equipment, coordination, balance)
  Interventions: Other: Clinical-neurological and neuropsychological tests; Diagnostic Test: Blood sampling; Other: Assessment of physical activity via fitness tracker/diary; Other: MRI-examinations
- control group (Other): continuation of physical activity as usual
  Interventions: Other: Clinical-neurological and neuropsychological tests; Diagnostic Test: Blood sampling; Other: Assessment of physical activity via fitness tracker/diary; Other: MRI-examinations

INTERVENTIONS:
Other: Clinical-neurological and neuropsychological tests — The tests include established standardized questionnaires and detailed clinical neuropsychological examinations (e.g., tests on cognition and perception). In order to avoid exercise effects in multiple examinations, so-called parallel procedures should be used.
Diagnostic Test: Blood sampling — Venous blood sampling (40 ml) is performed according to the usual criteria of sterile working at baseline and after intervention.
Other: Assessment of physical activity via fitness tracker/diary — All study participants, regardless of group classification, are randomly selected for a period of one week using Fitbit Charge 2® fitness trackers. The study participants are asked in this context to pursue their regular activity and to wear the bracelets for a week throughout. All study participants are asked to document their activities in a hand-written diary.
Other: MRI-examinations — Standard MRI-methods, Sodium MRI, Phosphor MRS, Wholebody-Fat-MRI

SUMMARY:
This study aims to gain a better understanding of metabolic early changes in neurodegenerative diseases, in order to enable new diagnostic and therapeutic approaches in the future. Further, it aims to identify specific movement-induced changes at the cerebral level, on cognition, on quality of life and physical fitness, and on serology parameters in neurodegenerative diseases.

In general, valid biomarkers are needed for early diagnosis and prediction of disease progression. It has been hypothesized that metabolic changes may precede structural changes and may be examined by intervention with exercise therapy. The non-invasive, in vivo characterization and diagnosis of such metabolic changes is therefore of paramount importance. In this line, this research project is focused on applying magnetic resonance imaging (MRI) based metabolic imaging techniques such as sodium MRI and phosphorus magnetic resonance spectroscopy (MRS) with standard structural and functional MRI methods, combined with exercise training, in order to detect biomarkers early in different stages of neurodegenerative diseases. Moreover, this project aims to examine the sensitivity of metabolic imaging with sodium and phosphorus sequences over classical MRI imaging with whole body fat sequences, in order to detect cerebral alterations.

At the end, the medical benefit of the planned project lies in the fact that the expected findings are groundbreaking for the understanding of the phenomenology and pathobiology of neurodegenerative diseases. This is the basis for the development of new methods for early diagnosis and individualized medicine with the optimization of future treatment options.

ELIGIBILITY:
Inclusion Criteria:

* prodromal or early symptomatic Alzheimer's disease according to the S3 guidelines of the German Society of Neurology in relation to the IWG-2 criteria for the definition of probable Alzheimer's disease
* Age between 50 and 80 years
* Mini Mental State Examination (MMSE)> 19 (screening at least 12 weeks before baseline visit)
* Cognitive ability to understand the task as well as regular participation in exercise program, based on assessment of the treating neurologist and / or neuropsychologist
* For antidementive or antidepressant medication, stable medication for at least 30 days
* No visual or auditory limitation preventing participation in cognitive and functional testing
* Interested in regular participation for 6 months, doing domestic exercises
* Presence of a written informed consent

Exclusion criteria:

* Heart attack or evidence of coronary heart disease (angina) in the last 2 years
* Severe systemic disease, which is expected to worsen during exercise
* Difficult to adjust diabetes mellitus II
* Difficult to set art. Hypertension in the last 6 months
* Severe psychiatric illness
* Severe orthopedic disease
* Alcohol and / or drug abuse in the last 2 years
* Chronic pain and / or musculoskeletal disease, which prevent regular physical activity
* Acute fracture or orthopedic injury last month
* cancer in the last 5 years (except basal cell and spinal cell carcinoma) Contraindications for MRI examination below 3 Tesla (for example, implantation of ferromagnetic parts) For study participants, the following measures must be observed due to the direct effects of the magnetic field, in particular the force exerted on para- or ferromagnetic bodies: Study participants with incorporated metallic implants are not admitted. Pregnancy or lactation, traumatic brain injury, neurological or psychiatric disorders (other than the neurological disease to be studied for patients), relevant and severe other medical conditions, e.g. metabolic, endocrinological or cardiac disorders, mental retardation, magnetic metal implants (also intrauterine spiral).

Furthermore, the spatial conditions in the magnet do not allow to examine persons with certain back complaints or a strong overweight. As a rule, a body mass index (BMI, weight [kg] / size2 [cm2]) of > 30 is the exclusion criterion. With regard to the participation in the exercise in advance with unclear suitability is a consultation with the attending family doctor regarding possible contraindications, which are a regular participation in a sports program in the way.

Specifically, as exclusion criteria count:

Diseases:

* epilepsy
* severe cardiac pre-existing conditions
* Musculoskeletal disorders that are contrary to regular exercise
* advanced osteoporosis
* Increased fall risk / imbalance
* Advanced Heart Failure, Shortness of Breath, Severe Pulmonary Disease, which are contrary to regular physical activity
* Diabetes mellitus prone to hypoglycaemia and hyperglycemia

Conditions:

* pregnancy
* Uncertain knowledge about possibly existing pregnancy

Contraceptives:

* Any type of intrauterine device
* Spiral made of copper Metal-containing implants or devices in / on the body (all non-metal implants / devices / patches will undergo a thorough examination based on the MRI Safety

Listing www.mrisafety.com):

* Pacemaker / implanted pacemaker wires
* Implanted defibrillator
* Drug pump / infusion device
* Stimulation device / electrodes

Non-MRI-compatible implants, for example, surgical screws, plates, nails, etc:

* vascular / lumen filters, wire rings, wire spirals, stents, vascular clips
* Artificial heart valve
* Transdermal patches
* epithesis (or partial epithesis)
* shunts, catheters, wire sutures

Metal in / on the body:

* Splinter / gunshot wounds
* Metal shards in the eye, even if everything was supposedly removed
* Piercing

Dental metals:

* Any type of implant in the jawbone area / dental implant older than 20 years
* No contraindications: Amalgam fillings, inlays, crowns, single crowned teeth as a denture base for a denture termed a telescopic denture, firmly screwed dentures

Additional:

* cochlear implant
* Ventilation Tubes
* tattoos / permanent make-up (only after the most exact examination and special approval see separate explanation)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Metabolic changes of the brain induced by intervention program | T1 (baseline), T3 (6 months, after intervention), T4 (optional, 1 year after intervention)
  Sodium MR Imaging
Metabolic changes of the brain induced by intervention program | T1 (baseline), T3 (6 months, after intervention), T4 (optional, 1 year after intervention)
  Phosphor MR Imaging
Structural changes of the brain induced by intervention program | T1 (baseline), T3 (6 months, after intervention), T4 (optional, 1 year after intervention)
  Standard MR Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Jörg B. Schulz, Prof. Dr., Study Director — Clinic for neurology University Hospital Aachen
Locations (1):
- RWTH Aachen University Hospital, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beckett MW, Ardern CI, Rotondi MA. A meta-analysis of prospective studies on the role of physical activity and the prevention of Alzheimer's disease in older adults. BMC Geriatr. 2015 Feb 11;15:9. doi: 10.1186/s12877-015-0007-2. PMID 25887627
- [Background] Bruggemann N, Hagenah J, Reetz K, Schmidt A, Kasten M, Buchmann I, Eckerle S, Bahre M, Munchau A, Djarmati A, van der Vegt J, Siebner H, Binkofski F, Ramirez A, Behrens MI, Klein C. Recessively inherited parkinsonism: effect of ATP13A2 mutations on the clinical and neuroimaging phenotype. Arch Neurol. 2010 Nov;67(11):1357-63. doi: 10.1001/archneurol.2010.281. PMID 21060012
- [Background] Diehl-Wiesenecker E, von Armin CA, Dupuis L, Muller HP, Ludolph AC, Kassubek J. Adipose Tissue Distribution in Patients with Alzheimer's Disease: A Whole Body MRI Case-Control Study. J Alzheimers Dis. 2015;48(3):825-32. doi: 10.3233/JAD-150426. PMID 26402111
- [Background] Hilker R, Klein C, Ghaemi M, Kis B, Strotmann T, Ozelius LJ, Lenz O, Vieregge P, Herholz K, Heiss WD, Pramstaller PP. Positron emission tomographic analysis of the nigrostriatal dopaminergic system in familial parkinsonism associated with mutations in the parkin gene. Ann Neurol. 2001 Mar;49(3):367-76. PMID 11261512
- [Background] Reetz K, Lencer R, Steinlechner S, Gaser C, Hagenah J, Buchel C, Petersen D, Kock N, Djarmati A, Siebner HR, Klein C, Binkofski F. Limbic and frontal cortical degeneration is associated with psychiatric symptoms in PINK1 mutation carriers. Biol Psychiatry. 2008 Aug 1;64(3):241-7. doi: 10.1016/j.biopsych.2007.12.010. Epub 2008 Feb 7. PMID 18261714
- [Background] Reetz K, Lencer R, Hagenah JM, Gaser C, Tadic V, Walter U, Wolters A, Steinlechner S, Zuhlke C, Brockmann K, Klein C, Rolfs A, Binkofski F. Structural changes associated with progression of motor deficits in spinocerebellar ataxia 17. Cerebellum. 2010 Jun;9(2):210-7. doi: 10.1007/s12311-009-0150-4. PMID 20016963
- [Background] Raj A, Kuceyeski A, Weiner M. A network diffusion model of disease progression in dementia. Neuron. 2012 Mar 22;73(6):1204-15. doi: 10.1016/j.neuron.2011.12.040. Epub 2012 Mar 21. PMID 22445347
- [Background] Warren JD, Rohrer JD, Hardy J. Disintegrating brain networks: from syndromes to molecular nexopathies. Neuron. 2012 Mar 22;73(6):1060-2. doi: 10.1016/j.neuron.2012.03.006. Epub 2012 Mar 21. PMID 22445334
- [Background] Zhou J, Gennatas ED, Kramer JH, Miller BL, Seeley WW. Predicting regional neurodegeneration from the healthy brain functional connectome. Neuron. 2012 Mar 22;73(6):1216-27. doi: 10.1016/j.neuron.2012.03.004. Epub 2012 Mar 21. PMID 22445348
- [Background] Jucker M, Walker LC. Pathogenic protein seeding in Alzheimer disease and other neurodegenerative disorders. Ann Neurol. 2011 Oct;70(4):532-40. doi: 10.1002/ana.22615. PMID 22028219